CLINICAL TRIAL: NCT07350421
Title: The Effectiveness of Inhaled Salbutamol in the Management of Transient Tachypnea of the Newborn(TTN)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TTN , newborn
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: TTN
Keywords: TTN; newboen
MeSH Terms: interventions — Albuterol; Saline Solution

STUDY DESIGN:
Intervention Model Description: The patient receives a single dose of inhaled salbutamol at a dose of 0.15 mg/kg mixed with 2 ml of 0.9% normal saline.
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A control group (Placebo Comparator): 2 ml of 0.9% saline solution for inhalation
  Interventions: Drug: Normal Saline
- B intervention group (Active Comparator): The patient receives a single dose of inhaled salbutamol at a dose of 0.15 mg/kg mixed with 2 ml of 0.9% normal saline.
  Interventions: Drug: Salbutamol (Albuterol)

INTERVENTIONS:
Drug: Salbutamol (Albuterol) — It belongs to a class of medications known as short-acting beta-2 adrenergic agonist.
  Arms: B intervention group
Drug: Normal Saline — normal saline by inhalation
  Arms: A control group

SUMMARY:
TTN is the most common respiratory disorder in the perinatal period, causing 40% of cases of respiratory distress after birth. Lung fluid absorption is initiated by beta-adrenergic agonists, such as endogenous steroids and Catecholamine, which increase during labor. Delayed absorption of fluid from the lungs is thought to be the primary mechanism of transient tachypnea of the newborn (TTN). The accumulation of fluid within the lungs impairs gas exchange, leading to increased respiratory effort. Tachypnea develops to compensate for this, and hypoxemia develops due to impaired alveolar ventilation . The main objective of the study:

To study the effectiveness of salbutamol in improving signs of respiratory distress according to the modified Downes score during the first 72 hours of life in infants with transient tachypnea of the newborn (TTN). Secondary objectives:

Duration of tachypnea (time to resolution of respiratory distress) Reducing the duration of the need for oxygen support Reducing the length of hospital stay

DETAILED DESCRIPTION:
Patients will be divided into two groups:

Intervention group B: receives a single dose of inhaled salbutamol at a dose of 0.15 mg/kg mixed with 2 ml of 0.9% normal saline.

Control group A: receives 2 ml of 0.9% normal saline. The study population consists of newborns born at Al-Ladhiqiyah University Hospital with a gestational age greater than 35 weeks who show signs of respiratory distress within the first 6 hours of birth.

ELIGIBILITY:
Inclusion Criteria:

Birth at the study hospital at a gestational age greater than 35 weeks. Clinical signs of TTN (tachypnea, retractions, grunting, nasal flaring) within the first 6 hours after birth.

-

Exclusion Criteria:

gestational age is 35 weeks or less. Meconium aspiration syndrome Pulmonary hypertension Congenital pneumonia and sepsis Congenital cardiovascular malformations Congenital thoracic and pulmonary malformations (diaphragmatic hernia, pulmonary hypoplasia, etc.)

-

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
study on the effectiveness of salbutamol in improving respiratory distress signs according to the modified Downes score during the first 72 hours of life in infants with TTN. | 72 hours
  Respiratory distress scores will be assessed using the modified Downes score ten minutes before the specified intervention is applied, and again at 6, 12, 24, 48, and 72 hours after the intervention begins.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Dayoub, PHD, Study Chair — Tishreen University
Locations (1):
- Latakia University, Latakia, Latakia Governorate, Syria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Danner D, Leder P. Role of an RNA cleavage/poly(A) addition site in the production of membrane-bound and secreted IgM mRNA. Proc Natl Acad Sci U S A. 1985 Dec;82(24):8658-62. doi: 10.1073/pnas.82.24.8658. PMID 3936040
- See also: Effects of Salbutamol on the Treatment of Transient Tachypnea of the Newborn — https://ijn.mums.ac.ir/article_11913_ad897e4c9f05fabcd12279661885daf5.pdf